CLINICAL TRIAL: NCT00387023
Title: Pilot Trial of Radioimmunotherapy With Yttrium 90-Labeled (90Y) Zevalin for Low-Grade Follicular Non-Hodgkin's Lymphoma or MALT of the Orbit/Conjunctiva
Brief Title: Radioimmunotherapy With 90Y Zevalin for Orbital Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0696
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-09

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Orbital Lymphoma; Rituximab; Rituxan; Zevalin; Ibritumomab tiuxetan; IDEC-Y2B8; Eye
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Orbital lymphoma | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zevalin + Rituximab (Experimental): Rituximab 250 mg/m^2 intravenous (IV) over 4-6 hours for 2 weeks, + Zevalin 5 millicurie (mCi)/kg IV over 30 minutes for 1 week, followed by 0.3 mCi/kg or 0.4 mCi/kg 90Y-Zevalin based on platelet counts for 1 week.
  Interventions: Drug: Rituximab; Drug: Zevalin

INTERVENTIONS:
Drug: Rituximab — 250 mg/m^2 IV over 4-6 hours for 2 weeks.
  Other Names: Rituxan
Drug: Zevalin — 5 mCi/kg IV over 30 minutes for 1 week, followed by 0.3 mCi/kg or 0.4 mCi/kg 90Y-Zevalin based on platelet counts for 1 week.
  Other Names: Ibritumomab tiuxetan; IDEC-Y2B8

SUMMARY:
Primary Objectives:

1. To evaluate the efficacy of Zevalin for the treatment of low-grade follicular Non-Hodgkin's lymphoma of the orbit or mucosa-associated lymphoid tissue (MALT) of conjunctiva using radiographic imaging, clinical examination (slit lamp biomicroscopy and external examination of the conjunctiva), and external photography whenever possible.
2. To establish the safety profile in this patient population using clinical examination including slit lamp biomicroscopy, and evaluation of the tear film with Schirmer's test.
3. To establish the dosimetry for Zevalin in the orbit in the first 3 patients who agree to undergo dosimetry.

DETAILED DESCRIPTION:
Rituximab and Zevalin are monoclonal antibodies that bind to lymphoma cells and cause cell death.

As is the case for all patients with orbital lymphoma, an orbital biopsy must be performed to confirm the diagnosis and status of the orbital lymphoma. The study doctors must first make sure that the disease has not spread too much and is not severe enough to require immediate treatment with chemotherapy before you can begin treatment on this study. You will have about 4 teaspoons of blood drawn. Women who are able to have children must have a negative blood or urine pregnancy test.

You will receive two injections of rituximab by vein over about 4 to 6 hours. This is followed by an infusion of Zevalin over about 30 minutes on the same day. Whole body images will be performed immediately and at 4-6, 24, 72, and 144 hours after receiving Zevalin. About 1 week later, you will receive a second infusion of rituximab and Zevalin.

You may be taken off the study if your orbital lymphoma does not respond within three months of receiving rituximab and Zevalin. Researchers will measure your response to therapy using magnetic Resonance imaging (MRI) of the orbit and an evaluation of the eye in the clinic. If you are taken off study, you will be given the option of receiving external beam radiation therapy as treatment for the disease.

Follow-up evaluations will be done every 3 months for 2 years and every 6 months for Years 3 and 4. This testing is considered standard of care and would include medical history, physical exam, blood tests, and urine tests. The status of the disease will be evaluated using CT scan or MRI of the orbit every 3 months for the first year and every 6 months for Years 2, 3, and 4. Blood tests (about 4 teaspoons each) will be every 3 months for the first year and may be continues every 3 to 6 month until they become negative or you start another anti-cancer therapy.

This is an investigational study. Zevalin and rituximab are both FDA approved but their use together in this study is investigational. A total of up to 12 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven diagnosis of low-grade Non-Hodgkin's follicular lymphoma of the orbit or MALT of the conjunctiva/orbit. The orbit/conjunctiva has to be the primary or predominant site of involvement or if there is a previous history of systemic involvement, the orbit/conjunctiva should be the only site of new recurrence.
2. No anti-cancer therapy for three weeks (six weeks if Rituximab, nitrosourea or Mitomycin C) prior to study initiation, and fully recovered from all toxicities associated with prior surgery, radiation treatments, chemotherapy, or immunotherapy
3. An Institutional Review Board (IRB)-approved signed informed consent
4. Age >18 years. This is justified since low-grade non-Hodgkin's lymphoma of the orbit is extremely rare to non-existent in the pediatric population
5. Expected survival of >3 months
6. Pre-study performance status of 0, 1, or 2 according to the WHO
7. Acceptable hematologic status within two weeks prior to patient registration, including: a) Absolute neutrophil count ([segmented neutrophils + bands] x total WBC)> 1500/mm3 b) Total lymphocyte count < 5,000/mm3 for patients with small lymphocytic lymphoma (IWFA) c) Platelet counts> 150,000/mm3, these patients will receive a dose of 0.4 mCi/kg of Zevalin d) Platelet counts from 100,00/mm3 to 149,000/mm3, these patients will receive a 0.3mCi/kg dose of Zevalin
8. Female patients who are not pregnant or lactating
9. Men and women of reproductive potential who are following accepted birth control methods (as determined by the treating physician, however abstinence is not an acceptable method)
10. Patients previously on Phase II drugs are eligible if no long-term toxicity is expected, and the patient has been off the drug for eight or more weeks with no significant post treatment toxicities observed
11. Patients determined to have less than 25% bone marrow involvement with lymphoma within six weeks of registration (based on a bone marrow biopsy). (This criteria must be strictly met for adequate patient safety.)

Exclusion Criteria:

1. Patients with impaired bone marrow reserve, as indicated by one or more of the following: a) Prior myeloablative therapies with autologous bone marrow transplantation (ABMT) or peripheral blood stem cell (PBSC) rescue b) Platelet count < than 100,000 cells/mm3 c) Hypocellular bone marrow (less than 15% cellularity) d) Marked reduction in bone marrow precursors of one or more cell lines (granulocytic, megakaryocytic, erythroid)
2. Prior radioimmunotherapy
3. Presence of central nervous system (CNS) lymphoma
4. Patients with HIV or AIDS-related lymphoma
5. Patients with small lymphocytic lymphoma (IWF A) - who have a total lymphocyte count > 5,000/mm3
6. Patients with pleural effusion
7. Patients with abnormal liver function: total bilirubin > 2.0 mg/dL
8. Patients with abnormal renal function: serum creatinine > 2.0 mg/dL
9. Patients who have received prior external beam radiation therapy to > 25% of active bone marrow (involved field or regional)
10. Patients who have received Granulocyte colony-stimulating factor (G-CSF or GM-CSF) therapy within two weeks prior to treatment
11. Serious nonmalignant disease or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives
12. Major surgery, other than diagnostic surgery, within four weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bita Esmaeli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment done at The University of Texas (UT) MD Anderson Cancer Center between August 2004 and November 2007.
Period: Overall Study
Arm/Group | Zevalin + Rituximab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Zevalin + Rituximab: Rituximab 250 mg/m^2 intravenous (IV) over 4-6 hours for 2 weeks, + Zevalin 5 mCi/kg IV over 30 minutes for 1 week, followed by 0.3 mCi/kg or 0.4 mCi/kg 90Y-Zevalin based on platelet counts for 1 week.
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 12
Age Continuous [Median (Full Range); unit: years] | 60 [22 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: Tumor response to therapy measured by tumor size as measured radiographically at baseline and at three months from baseline. Tumor response classified as complete response (CR) or partial response (PR), or stable disease (SD), or progressive disease (PD) using International Workshop Standardized Response Criteria (IWC) for Non-Hodgkin's Lymphomas. If the orbital/ocular adnexal lymphoma was not evaluable radiographically, clinical evaluation using slit lamp biomicroscopy was used to assess PR or CR.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 12
participants
  CR | 10
  PR | 2

ADVERSE EVENTS:
Time Frame: 7 years and 2 months
Arm/Group | Zevalin + Rituximab
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zevalin + Rituximab (N=12)
Transient Pancytopenia (Blood and lymphatic system disorders) | 12
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 8
Increased Bruisability (General disorders) | 7
Joint and Muscle Pain (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Headache (General disorders) | 3
Fever (Infections and infestations) | 1
Dizziness (General disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No